CLINICAL TRIAL: NCT05749445
Title: Appropriate Evaluation of Antiviral Therapy With Nirmatrelvir-ritonavir in Hospitalized Patients: a Multicenter Retrospective Study in China
Brief Title: Appropriate Evaluation of Antiviral Therapy With Nirmatrelvir-ritonavir in Hospitalized Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Hangzhou Cancer Hospital (Other); First People's Hospital of Lin'an District (Unknown); First People's Hospital of Yuhang District (Unknown)
Responsible Party: Sponsor
Other Study IDs: AEATN
Record Dates: First submitted 2023-02-16; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Hospitalized Patients
MeSH Terms: interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nirmatrelvir-Ritonavir: Hospitalized patients receiving at least one dose Nirmatrelvir-Ritonavir
  Interventions: Drug: Nirmatrelvir-Ritonavir

INTERVENTIONS:
Drug: Nirmatrelvir-Ritonavir — Nirmatrelvir-Ritonavir
  Other Names: PAXLOVID

SUMMARY:
The primary objective of the study was to assess the appropriateness of antiviral therapy with nirmatrelvir-ritonavir in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients receiving at least one dose nirmatrelvir-ritonavir

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized patients receiving at least one dose nirmatrelvir-ritonavir
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The prevalence of inappropriate use of nirmatrelvir-ritonavir | baseline
  Four aspects were evaluated to identify the rationality of prescribing NMVr, including indication, administration (dose, timing, and duration), contraindications, and drug-drug interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Changcheng Shi, Principal Investigator — First People's Hospital of Hangzhou
Locations (1):
- Changcheng Shi, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamb YN. Nirmatrelvir Plus Ritonavir: First Approval. Drugs. 2022 Apr;82(5):585-591. doi: 10.1007/s40265-022-01692-5. PMID 35305258
- [Background] Akinosoglou K, Schinas G, Gogos C. Oral Antiviral Treatment for COVID-19: A Comprehensive Review on Nirmatrelvir/Ritonavir. Viruses. 2022 Nov 17;14(11):2540. doi: 10.3390/v14112540. PMID 36423149
- See also: COVID-19 Drug Interactions — http://www.covid19-druginteractions.org
- See also: Fact sheet for healthcare providers: Emergency use authorization for Paxlovid — http://www.fda.gov/media/155050/download